CLINICAL TRIAL: NCT03650452
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-935 (OV935) as an Adjunctive Therapy in Pediatric Patients With Developmental and/or Epileptic Encephalopathies
Brief Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-935 (OV935) as an Adjunctive Therapy in Pediatric Participants With Developmental and/or Epileptic Encephalopathies
Acronym: ELEKTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Healx AI (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-935-2002; U1111-1206-5522 (Other: World Health Organization); 2018-002484-25 (EudraCT Number)
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Epilepsy; Dravet Syndrome; Lennox-Gastaut Syndrome
Keywords: Drug Therapy; Brain Diseases; Central Nervous System Diseases; Tuberous Sclerosis; CDKL5 deficiency disorder; Dup15Q syndrome; Anoxic brain injury; Infantile spams; West syndrome; Cortical dysplasia; SCN1A; OV-935; Cholesterol 24S-hydroxylase inhibitor; Seizure; Anti-epileptic drug; Anticonvulsants; Nervous System Diseases; Drop seizure; Atonic seizure
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Lennox Gastaut Syndrome; Brain Diseases; Central Nervous System Diseases; Tuberous Sclerosis; CDKL5 deficiency disorder; Hypoxia-Ischemia, Brain; Spasms, Infantile; Malformations of Cortical Development; Seizures; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): TAK-935 placebo-matching tablets, orally or via gastrostomy tube (G-tube)/percutaneous endoscopic gastrostomy (PEG), twice a day (BID) up to Week 20.
  Interventions: Drug: Placebo
- TAK-935 (Experimental): TAK-935 tablets orally or via G-tube/PEG tube, BID. Participants weighing <60 kg received total daily dose of study drug calculated based on body weight. Participants weighing ≥60 kg at Baseline, were administered with 200 mg/day followed by 400 mg/day, then 600 mg/day, up to Week 20.
  Interventions: Drug: TAK-935

INTERVENTIONS:
Drug: TAK-935 — TAK-935 tablets or mini-tablets.
  Arms: TAK-935
Drug: Placebo — TAK-935 placebo-matching tablets or mini-tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect on the frequency of all seizures (convulsive and drop) in participants treated with TAK-935 compared to placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-935 (OV935). This randomized, double-blind study will assess the effects of TAK-935 (OV935), compared to placebo, on efficacy, safety, and tolerability in pediatric participants with Dravet syndrome (DS) or Lennox Gastaut syndrome (LGS). This multi-center trial will be conducted worldwide and will enroll approximately 126 participants.

Participants will be randomized based on their diagnosis in 2 categories; DS or LGS. The study will consist of 2 periods: Screening Period and Treatment Period. The overall duration of Treatment Period is up to 20 weeks including 8-week Dose Optimization Period and 12-week Maintenance Period. The overall time to participants in this study is approximately 30 weeks.

Participants completing this study will have an option to enroll in the open-label extension study, under a separate protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged greater than or equal to (>=) 2 and less than or equal to (<=) 17 years
2. Clinical diagnosis of DS or LGS
3. Weight of >=10 kilogram (kg) at the Screening visit
4. Currently taking 1 to 4 anti-epileptic drugs (AEDs) at a stable dose
5. Failed to become and remain seizure free with trials of at least 2 AEDs

Exclusion Criteria:

1. Has been admitted to a medical facility and intubated for treatment of status epilepticus 2 or more times in the 3 months immediately prior to the screening visit
2. Non-epileptic events that cannot be reliably distinguished from epileptic seizures
3. Participation in a clinical study involving another study drug in the previous month

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (44):
- United States (15):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Nicklaus Children's Hospital, Miami, Florida
  - Pediatric Neurology PA, Orlando, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Center for Rare Neurological Diseases, Norcross, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Children's Hospital at Saint Peter's University Hospital, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Cook Children's Medical Center, Fort Worth, Texas
- Australia (2):
  - Monash Children's Hospital, Clayton, Victoria
  - Austin Hospital, Heidelberg West, Victoria
- Hospital For Sick Children, Toronto, Ontario, Canada
- China (6):
  - Peking University First Hospital, Beijing
  - Capital Medical University (CMU) - Beijing Children's Hospital, Beijing
  - Beijing Children's Hospital,Capital Medical University, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Children's Hospital of Fudan University, Shanghai
  - Shenzhen Children's Hospital, Shenzhen
- Israel (7):
  - Sheba Medical Center-PPDS, Tel Litwinsky, Ramat Gan
  - Soroka University Medical Centre, Bear Sheva
  - Bnai Zion Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Schneider Childrens Medical Center of Israel, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Poland (6):
  - Szpital Kliniczny im. H.Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan, Greater Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne - PPDS, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Plejady, Krakow
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny w Warszawie, Warsaw
  - Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw
  - NZOZ Centrum Neurologii Dzieciecej i Leczenia Padaczki, Kielce, Świętokrzyskie Voivodeship
- Portugal (3):
  - Centro Hospitalar Lisboa Central- Hospital Dona Estefania, Lisbon
  - Centro Hospitalar Lisboa Norte, E.P.E. Hospital de Santa Maria, Lisbon
  - Largo da Maternidade de Julio DinisCentro Materno Infantil do Norte, Porto
- Spain (4):
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Vithas La Salud, Granada
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hahn CD, Jiang Y, Villanueva V, Zolnowska M, Arkilo D, Hsiao S, Asgharnejad M, Dlugos D. A phase 2, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of soticlestat as adjunctive therapy in pediatric patients with Dravet syndrome or Lennox-Gastaut syndrome (ELEKTRA). Epilepsia. 2022 Oct;63(10):2671-2683. doi: 10.1111/epi.17367. Epub 2022 Aug 4. PMID 35841234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 45 investigative sites globally from 8 August 2018 to 20 July 2020.
Pre-assignment Details: Participants with a diagnosis of Dravet syndrome (DS) or Lennox-Gastaut syndrome (LGS) were enrolled and randomized in a 1:1 ratio to double-blind treatment with TAK-935 or matching placebo for up to the 20-week Treatment Period (8-week Dose Optimization Period and 12-week Maintenance Period).
Period: Overall Study
Arm/Group | Placebo | TAK-935
Started | 70 | 71
Completed | 60 | 66
Not Completed | 10 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 3 | 1
Not completed — Adverse Event | 3 | 4
Not completed — Early Withdrawal from Study Treatment | 3 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set included all participants who were randomized into the study.
Groups:
- Placebo: TAK-935 placebo-matching tablets, orally or via G-tube/PEG, BID up to Week 20.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-935 | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (3.93) | 9.6 (4.14) | 9.5 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 42 | 49 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 60 | 60 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 22 | 22 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 47 | 49 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 2 | 2 | 4
  Canada | 3 | 3 | 6
  China | 20 | 21 | 41
  Spain | 11 | 8 | 19
  Israel | 5 | 4 | 9
  Poland | 12 | 17 | 29
  Portugal | 2 | 3 | 5
  United States | 15 | 13 | 28
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed are the number of participants with data available for height at Baseline.
  cm
    number analyzed (Participants) | 68 | 71 | 139
    (all) | 132.4 (20.34) | 134.7 (21.34) | 133.6 (20.81)
Weight [Mean (Standard Deviation); unit: kg] | 32.8 (15.98) | 33.3 (15.11) | 33.0 (15.49)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2)] — BMI= weight (kg)/height (m^2). Population: Number analyzed are the number of participants with data available for BMI at Baseline.
  (kg/m^2)
    number analyzed (Participants) | 68 | 71 | 139
    (all) | 17.63 (4.378) | 17.43 (4.048) | 17.53 (4.198)
Clinical Global Impression of Severity (CGI-S) Responses of Investigator [Mean (Full Range); unit: score on a scale] — The CGI-Severity (CGI-S) focuses on clinicians' observations of the participant's cognitive, functional, and behavioral performance since the beginning of the study. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill participants). Population: Efficacy Analysis Set included all mITT participants whose efficacy assessments were compliant with Protocol Amendment 2.
  score on a scale
    number analyzed (Participants) | 59 | 64 | 123
    (all) | 4.8 [3 to 7] | 4.5 [2 to 7] | 4.65 [2 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Seizure Frequency Per 28 Days During the Maintenance Period
Description: Seizure frequency per 28 days is defined as total number of seizures (convulsive seizures for DS, drop seizures for LGS) reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent change from Baseline is defined as (frequency of seizures per 28 days during maintenance period - frequency of seizures per 28 days at baseline) divided by frequency of seizures per 28 days at baseline multiplied by 100. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline; Maintenance Period: Weeks 9 to 20
Population: Efficacy Analysis Set included all Modified Intent-to-Treat (mITT) participants whose efficacy assessments were compliant with Protocol Amendment 2. Overall number analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 56 | 64
percent change | 3.11 [-78.8 to 163.0] | -27.76 [-100.0 to 160.6]
Statistical Analysis 1: Comparison: Placebo vs TAK-935; Test type: Superiority; p = 0.0007, Ranked ANCOVA — The p-value is 2-sided and it is for the difference of percent change from baseline between TAK-935 and Placebo were computed using Rank Transformed Analysis of Covariance (ANCOVA) adjusting for baseline seizure frequency and indication; Hodges-Lehmann Estimation = -30.48, 95% CI 2-sided [-46.99 to -13.19] — The location shift (TAK-935 - Placebo) and Asymptotic 95% confidence interval between TAK-935 and Placebo (TAK-935 - Placebo) were based on Hodges-Lehmann Estimation from un-adjusted rank statistics

2. Secondary Outcome: Percent Change From Baseline in Seizure Frequency Per 28 Days During the Treatment Period
Description: Seizure Frequency per 28 days is defined as total number of Seizures reported (convulsive seizures for DS, drop seizures for LGS) during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent Change from Baseline is defined as (frequency of seizures per 28 days during treatment period - frequency of seizures per 28 days at baseline) divided by frequency of seizures per 28 days at baseline multiplied by 100. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline; Treatment Period: Weeks 0 to 20
Population: Efficacy Analysis Set included all mITT participants whose efficacy assessments were compliant with Protocol Amendment 2.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 59 | 64
percent change | 0.75 [-60.1 to 437.8] | -30.05 [-100.0 to 347.5]
Statistical Analysis 1: Comparison: Placebo vs TAK-935; Test type: Superiority; p = 0.0024, Ranked ANCOVA — The p-value is 2-sided and it is for the difference of percent change from baseline between TAK-935 and Placebo were computed using Rank Transformed ANCOVA adjusting for baseline seizure frequency and indication; Hodges-Lehmann Estimate = -25.93, 95% CI 2-sided [-43.96 to -10.69] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Change From Baseline in Convulsive Seizure Frequency Per 28 Days in Participants With Dravet Syndrome Stratum During the Maintenance Period
Description: Convulsive seizure frequency per 28 days is defined as total number of convulsive seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent Change from Baseline (%) is defined as [(Maintenance Period Convulsive Seizure Frequency - Baseline Period Convulsive Seizure Frequency) divided by Baseline Convulsive Seizure Frequency] multiplied by 100. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline; Maintenance Period: Weeks 9 to 20
Population: Efficacy Analysis Set included all mITT participants whose efficacy assessments were compliant with Protocol Amendment 2. Overall number analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 21 | 24
percent change | 9.38 [-47.3 to 153.5] | -36.50 [-100.0 to 84.1]
Statistical Analysis 1: Comparison: Placebo vs TAK-935; Test type: Superiority; p = 0.0001, Ranked ANCOVA — The p-value is 2-sided and it is for the difference of percent change from baseline between TAK-935 and Placebo were computed using Rank Transformed ANCOVA adjusting for baseline seizure frequency; Hodges-Lehmann Estimate = -50.00, 95% CI 2-sided [-75.03 to -25.09] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Change From Baseline in Drop Seizure Frequency Per 28 Days in Participants With the Lennox-Gastaut Syndrome (LGS) Stratum During the Maintenance Period
Description: Drop seizure frequency per 28 days is defined as total number of drop seizures reported during the period divided by number of days during the period seizures were assessed multiplied by 28. Percent Change from Baseline (%) is defined as [(Maintenance Period Drop Seizure Frequency - Baseline Period Drop Seizure Frequency) divided by Baseline Drop Seizure Frequency] multiplied by 100. Negative percent change from Baseline indicates improvement.
Time Frame: Baseline; Maintenance Period: Weeks 9 to 20
Population: as for outcome 3
Measure: Median (Full Range); unit: percent change
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 35 | 40
percent change | -1.90 [-78.8 to 163.0] | -18.46 [-100.0 to 160.6]
Statistical Analysis 1: Comparison: Placebo vs TAK-935; Test type: Superiority; p = 0.1470, Ranked ANCOVA — [p-value comment as in outcome 3, analysis 1]; Hodges-Lehmann Estimate = -16.22, 95% CI 2-sided [-39.50 to 4.49] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With LGS Stratum Considered Treatment Responders Throughout the Maintenance Period
Description: Responders are defined as having over 50% drop seizure reduction compared to Baseline. Percent Reduction from Baseline (%) is defined as [(Maintenance Period Drop Seizure Frequency - Baseline Period Drop Seizure Frequency) divided by Baseline Drop Seizure Frequency] multiplied by 100. Data is reported as reduction of 25%, 50%, 75% and 100% or more in drop seizures from Baseline.
Time Frame: Maintenance Period: Weeks 9 to 20
Population: Efficacy Analysis Set included all mITT participants whose efficacy assessments were compliant with Protocol Amendment 2. Only participants with LGS stratum indication were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 37 | 40
percentage of participants
  Reduction of 25% or More in Drop Seizures from Baseline | 29.7 [15.9 to 47.0] | 42.5 [27.0 to 59.1]
  Reduction of 50% or More in Drop Seizures from Baseline | 16.2 [6.2 to 32.0] | 27.5 [14.6 to 43.9]
  Reduction of 75% or More in Drop Seizures from Baseline | 2.7 [0.1 to 14.2] | 10.0 [2.8 to 23.7]
  Reduction of 100% in Drop Seizures from Baseline | 0 [0.0 to 9.5] | 5.0 [0.6 to 16.9]

6. Secondary Outcome: Percentage of Participants With Dravet Syndrome Stratum Considered Treatment Responders Throughout the Maintenance Period
Description: Responders are defined as having over 50% convulsive seizure reduction compared to Baseline. Percent Reduction from Baseline (%) is defined as [(Maintenance Period Convulsive Seizure Frequency - Baseline Period Convulsive Seizure Frequency) divided by Baseline Convulsive Seizure Frequency] multiplied by 100. Data is reported as reduction of 25%, 50%, 75% and 100% or more in drop seizures from Baseline.
Time Frame: Maintenance Period: Weeks 9 to 20
Population: Efficacy Analysis Set included all mITT participants whose efficacy assessments were compliant with Protocol Amendment 2. Only participants with Dravet syndrome stratum indication were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 22 | 24
percentage of participants
  Reduction of 25% or More in Convulsive Seizures from Baseline | 13.6 [2.9 to 34.9] | 66.7 [44.7 to 84.4]
  Reduction of 50% or More in Convulsive Seizures from Baseline | 0 [0.0 to 15.4] | 41.7 [22.1 to 63.4]
  Reduction of 75% or More in Convulsive Seizures from Baseline | 0 [0.0 to 15.4] | 20.8 [7.1 to 42.2]
  Reduction of 100% in Convulsive Seizures from Baseline | 0 [0.0 to 15.4] | 8.3 [1.0 to 27.0]

7. Secondary Outcome: Change From Baseline in Clinician's Clinical Global Impression of Severity (CGI-S) Responses of Investigator Reported Impression of Efficacy and Tolerability of Study Drug
Description: The CGI-Severity (CGI-S) focuses on clinicians' observations of the participant's cognitive, functional, and behavioral performance since the beginning of the study. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill participants). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 20
Population: as for outcome 3
Measure: Least Squares Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 49 | 58
score on scale | -0.3 (0.15) | -0.2 (0.14)
Statistical Analysis 1: Comparison: Placebo vs TAK-935; Test type: Superiority; p = 0.6829, Mixed-Model Repeated Measure (MMRM) — The p-value is 2-sided and it is for the difference (TAK-935 - Placebo) of change from baseline between TAK-935 and Placebo was computed using MMRM; Least Square (LS) Mean = 0.1, 95% CI 2-sided [-0.32 to 0.49], Standard Deviation 0.21 — The MMRM model included treatment and visit as factors along with treatment*visit interaction and baseline score as a covariate; and visit as repeated measure

8. Secondary Outcome: Percentage of Participants With Clinical Global Impression of Change (CGI-C) Responses as Per the Investigator Reported Impression of Efficacy and Tolerability TAK-935
Description: CGI-Change (CGI-C) treatment response ratings should take account of both therapeutic efficacy and treatment-related AEs. Each component of the CGI is rated separately; the instrument does not yield a global score. The CGI-C is rated on a 7-point scale, where, 0 = Marked improvement and no side-effects, 1 = Marked improvement and minimal side-effects, 2 = No Change, 3 = Minimal improvement and marked side-effects and 4 = Unchanged or worse and side-effects outweigh the therapeutic effect. Lower scores indicated improvement.
Time Frame: Week 20
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 49 | 58
percentage of participants
  Week 20, Score 0 | 12.2 | 17.2
  Week 20, Score 1 | 2.0 | 15.5
  Week 20, Score 2 | 85.7 | 65.5
  Week 20, Score 3 | 0 | 0
  Week 20, Score 4 | 0 | 1.7

9. Secondary Outcome: Percentage of Participants With Caregiver Global Impression of Change (Care GI-C) Responses as Per the Parent/Family Reported Impression of Efficacy and Tolerability of TAK-935
Description: The Care GI-C is rated on a 7-point scale, with the severity of illness scale where, 1 = Very much improved, 2 = Much improved, 3 = Slightly improved, 4 = No change, 5 = Slightly worse, 6 = Much worse and 7 = Very much worse. Lower scores indicated improvement.
Time Frame: Week 20
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 49 | 58
percentage of participants
  Week 20, Score 1 | 2.0 | 13.8
  Week 20, Score 2 | 12.2 | 10.3
  Week 20, Score 3 | 18.4 | 32.8
  Week 20, Score 4 | 55.1 | 37.9
  Week 20, Score 5 | 8.2 | 3.4
  Week 20, Score 6 | 4.1 | 1.7
  Week 20, Score 7 | 0 | 0

10. Secondary Outcome: Change From Baseline in Plasma 24S-Hydroxycholesterol (24HC) Levels in Participants Treated With TAK-935 as an Adjunctive Therapy
Description: A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Efficacy Analysis Set included all mITT participants whose efficacy assessments were compliant with Protocol Amendment 2, with available data. Number analyzed is the number of participants with Baseline and Week 24 data available for analyses.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 57 | 61
mg/dL
  Baseline | 102.77 (50.385) | 102.20 (62.332)
  Change from Baseline at Week 24: number analyzed (Participants) | 0 | 1
  Change from Baseline at Week 24 |  | -0.10 (NA) — Standard deviation was not estimable for 1 participant.

11. Secondary Outcome: Change From Baseline in Seizure Frequency in Participants Treated With TAK-935 as an Adjunctive Therapy
Description: Seizure frequency was based on convulsive seizures for the participants in the Dravet Syndrome Indication and Drop Seizures for the participants in the LGS Indication. Seizure frequency per 28 days = (total number of seizures reported during the period) / (number of days during the period seizures were assessed) * 28. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 20
Population: as for outcome 10
Measure: Median (Full Range); unit: seizures per 28 days
Arm/Group | Placebo | TAK-935
Number analyzed (Participants) | 57 | 61
seizures per 28 days
  Baseline | 31.00 [3.1 to 1040.1] | 32.12 [2.6 to 5187.7]
  Change from Baseline at Week 20: number analyzed (Participants) | 33 | 40
  Change from Baseline at Week 20 | 0.30 [-84.9 to 520.4] | -6.29 [-1024.3 to 77.7]

ADVERSE EVENTS:
Time Frame: From the first dose to 30 days post-last dose of study treatment (Up to 24 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-935
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71
Serious Adverse Events (participants affected / at risk) | 13/70 | 11/71
Other Adverse Events (participants affected / at risk) | 52/70 | 55/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=70) | TAK-935 (N=71)
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 2 | 2
Seizure cluster (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 1
Tonic convulsion (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=70) | TAK-935 (N=71)
Nasopharyngitis (Infections and infestations) | 6 | 6
Upper respiratory tract infection (Infections and infestations) | 10 | 12
Pyrexia (General disorders) | 8 | 11
Seizure (Nervous system disorders) | 7 | 4
Somnolence (Nervous system disorders) | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 4 | 6
Decreased appetite (Metabolism and nutrition disorders) | 5 | 6
Basophilia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 3
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Amblyopia (Eye disorders) | 1 | 0
Blepharitis (Eye disorders) | 1 | 0
Excessive eye blinking (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Periorbital swelling (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Decreased activity (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 4
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 1
Gingival abscess (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 2
Laryngitis (Infections and infestations) | 1 | 1
Nail infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 3 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tonsillitis bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 3 | 2
Benzodiazepine drug level increased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 3 | 0
Blood calcium decreased (Investigations) | 0 | 1
Blood pressure diastolic increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
Drug level increased (Investigations) | 0 | 1
Electrocardiogram P wave abnormal (Investigations) | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Electrocardiogram repolarisation abnormality (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Nitrite urine present (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Protein urine present (Investigations) | 1 | 2
Prothrombin time prolonged (Investigations) | 0 | 1
Red blood cells urine (Investigations) | 1 | 0
Urine output decreased (Investigations) | 0 | 1
Vitamin D decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cerebellar ataxia (Nervous system disorders) | 0 | 1
Change in seizure presentation (Nervous system disorders) | 1 | 0
Chorea (Nervous system disorders) | 0 | 1
Clonic convulsion (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 1 | 3
Epilepsy (Nervous system disorders) | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 0 | 3
Hypersomnia (Nervous system disorders) | 1 | 2
Hypotonia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 5
Myoclonic epilepsy (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 2 | 1
Poor quality sleep (Nervous system disorders) | 0 | 1
Seizure cluster (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 3
Affect lability (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Apathy (Psychiatric disorders) | 0 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 0
Defiant behaviour (Psychiatric disorders) | 0 | 1
Impulsive behaviour (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1
Irritability (Psychiatric disorders) | 2 | 4
Middle insomnia (Psychiatric disorders) | 1 | 1
Negativism (Psychiatric disorders) | 0 | 1
Poverty of speech (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Hypercalciuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Erection increased (Reproductive system and breast disorders) | 1 | 0
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Pallor (Vascular disorders) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Tonic convulsion (Nervous system disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT03650452/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT03650452/SAP_001.pdf